CLINICAL TRIAL: NCT05989477
Title: At-home Breast Oncology Care Delivered With E-health Solutions The ABODE Study
Brief Title: At-home Breast Oncology Care Delivered With E-health Solutions
Acronym: ABODE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-6232
Record Dates: First submitted 2023-06-14; First posted 2023-08-14 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Patient Engagement; Patient Activation; Patient Reported Outcome Measures
Keywords: e-Health; m-Health; Mobile Application; Psychosocial Oncology; Survivorship; Breast Cancer
MeSH Terms: conditions — Patient Participation; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The intervention group (n=100) will receive access to the app in addition to standard care for 13 months following their diagnosis. The control group (n=100) will have standard care.
Masking Description: After randomization patients will be told what experimental arm they are in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): The control arm will receive standard treatment.
- Interventional Arm (Experimental): Individuals within the intervention will receive standard care and access to the Breast Cancer Treatment Application (BCTA) for 13 months.
  Interventions: Other: At-home Breast Oncology care Delivered with E-health solutions - ABODE

INTERVENTIONS:
Other: At-home Breast Oncology care Delivered with E-health solutions - ABODE — The development and implementation of the Breast Cancer Treatment Application (BCTA) will facilitate a secure approach to virtual care for Breast Cancer patients, provide patient specific treatment education and facilitate evaluation of Patient Reported Outcome Measures.
  Arms: Interventional Arm

SUMMARY:
The COVID-19 pandemic has significantly impacted healthcare service delivery, highlighting the need for high quality virtual patient care. Our team has developed a multi-dimensional remote eHealth solution for newly diagnosed breast cancer patients and their practitioners to use during the diagnostic and follow-up period. The ABODE study involved development of a Breast Cancer Treatment Application (app) which will facilitate virtual consultations, deliver patient education material, and collect patient reported outcome measures (PROMs). Using a randomized controlled trial design, the team will evaluate a variety of outcomes for breast cancer patients who will use the app throughout their diagnosis and treatment period.

Primary Objective: To compare changes in patient activation (assessed by PAM-13) over 1 year among newly diagnosed breast cancer patients between those using the app and those receiving standard care.

Secondary Objectives:

1. Compare additional PROMs between the standard care and intervention groups
2. Describe health service outcomes among app users
3. Explore end-user experience of using the app
4. Measure activity levels using wearable devices

DETAILED DESCRIPTION:
To measure the effect of the app compared to the standard care approach, the study team will conduct a randomized controlled trial of 200 newly diagnosed breast cancer patients seen at a tertiary care cancer centre in Ontario, Canada. The intervention group (n=100) will receive access to the app in addition to standard care for 13 months following their diagnosis. The control group (n=100) will have standard care. Both arms will be provided with a Fitbit wearable device.

The PAM-13 scale assesses patient activation, defined as the knowledge and confidence a patient has in self- management of one's health. Research team will test whether use of the app improves PAM-13 scores at the 12-month follow-up.

Additionally, secondary outcomes will be assessed with data from additional patient-reported outcome measures (PROMs), chart review, hospital administrative databases, and Fitbits. All participants will complete PROMs at baseline, 6- and 12- months post diagnosis via REDCap survey links sent through email. The intervention group will have access to the app for 13 months following randomization.

ELIGIBILITY:
Inclusion Criteria:

* Females (assigned female at birth)*
* Diagnosed with first, primary invasive BC
* Must have surgery as their first step in treatment pathway
* Age≥18
* Access to an electronic device with connection to the internet
* A valid email address
* Can communicate in English *Since BC risk is sex-related and based on physiological values, our inclusion criteria are based on sex (not gender)

Exclusion criteria:

* Males (assigned male at birth), as BC surgical treatment options and experiences are different
* Diagnosed with non-operable breast cancer
* Stage 4/metastatic (whether determined at diagnosis or during surgery)
* Those with hearing or visual challenges
* Neo-adjuvant chemotherapy
* Should not be enrolled in any other UHN study using an e-Health application
* Breast cancer surgery is scheduled for less 5 business days after enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-22 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | At baseline, 6 months and 12 months after enrollment
  To compare changes in patient activation (assessed by Patient Activation Measure -13) over 1 year among newly diagnosed breast cancer patients between those using the Breast Cancer Treatment Application (BCTA) and those receiving standard care.
  Difference in Patient Activation Measure (PAM) scores between pre/post intervention. PAM includes 13 questions, each with 4 response options, summed on a 0-100 scale, with higher scores indicating higher activation level.
  Patient activation is defined as the knowledge, skills, and confidence a person has in managing their health and care. Studies have shown that higher patient activation is associated with improved health related quality of life (HRQoL) and lower health care utilization.

SECONDARY OUTCOMES:
PROM 1: Impact of Events Scale - Revised (IES-R) | At baseline, 6 and 12 months after diagnosis
  Number of participants with PTSD symptoms, such as distress in regards to their Breast Cancer diagnosis and treatment as assessed by IES-R.
  Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). The IES-R yields a total score (ranging from 0 to 88); higher scores mean worse symptoms.
PROM 2: Generalized Anxiety Disorder (GAD-7) | At baseline, 6 and 12 months after diagnosis
  Number of participant with generalized anxiety around their breast cancer diagnosis and treatment assessed by GAD-7.
  The GAD-7 is a 7-item scale used to measure or assess the severity of generalized anxiety disorder based on symptoms.
PROM 3: European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire (EORTC QLQ-C30) | At baseline, 6-months and 12-months post-diagnosis
  Number of participants with changes in their physical, psychological and social functions during and after their diagnosis and surgery, assessed by the EORTC QLQ-C30.
  The EORTC Core Questionnaire (QLQ-C30) includes six clearly distinguishable functioning scales that have been thoroughly tested and validated on an international level and that are available in 110 different language versions. About the functional scale and the global health status, the higher the total score, the better the quality of life; the lower the score in the symptom scale, the better the quality of life.
PROM 4: European Organisation for Research and Treatment of Cancer - Breast Cancer-Specific Quality of Life Questionnaire (EORTC QLQ-BR23) | At baseline, 6-months and 12-months after enrollment
  Number of participants with changes in their quality of life after their breast cancer diagnosis and treatment journey assessed by the EORTC QLQ-BR23.
  The survey includes functional scales (body image, sexual functioning, sexual enjoyment, and future perspective) and single item symptoms scales (systemic therapy side effects, breast symptoms, arm symptoms, and upset by hair loss). Questions used 4-point Likert scale (1 'Not at All' to 4 'Very Much'). Scores average and transformed to 0-100 scale. High score for functional scale=high/healthy level of functioning. High score for single item=high level of symptomatology/problems.
PROM 5: Self-Identification Survey | At baseline
  Number of participants and their reported identities assessed by the self-identification survey.
PROM 6: European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire INFO 25 (EORTC QLQ-INFO 25). | 9-months post-diagnosis
  Number of participants and their satisfaction with information provided about treatment received assessed by the EORTC QLQ-INFO25.
  The provisional 25-item information questionnaire is Questions used 4-point Likert scale (1 'Not at All' to 4 'Very Much'). Scores average and transformed to 0-100 scale. High score for functional scale=higher satisfaction with provided treatment information.
PROM 7: The Health Information Questionnaire (heiQ) | At baseline, 9 months post-diagnosis
  Number of participants and how comfortable they are with the patient educational programs provided throughout the patient's treatment journey, assessed by the heiQ at the beginning and 9 months post diagnosis.
  heiQ is a validated, self-reported instrument with 8 domains to comprehensively evaluate patient education program and self-management intervention. Each domain score ranges from 1 to 4; a higher score indicates better outcome.
PROM 8: Clinical Evaluation Questionnaire - INS (CEQ-INS) | 6 and 12 months post-diagnosis
  Number of participants and their experience of cancer care in teams of their receipt of useful and relevant information about cancer, assistance with service navigation, and support from their care team examined with the CEQ-INS half way and end of the study.
  CEQ-INS is a self-reported instrument with questions used 4-point Likert scale (1 'Not at All' to 4 'Very Much'). Higher scores correlate with higher patient satisfaction with the information and support provided from their care team.
PROM 9: Other Health App Questionnaire (OHA) | 6 and 12 months post-diagnosis
  Number of participants and how frequently they use other e-health applications assessed by the OHA.
  The OHA is a self reported questionnaire with an array question (yes, no, unsure) regarding the participants involvement with other e-health applications.
PROM 10: The Duke Activity Status Index (DASI) | Baseline
  Number of participants and their functional capacity evaluated by the DASI at the beginning of the study.
  The Duke Activity Status Index (DASI) is a 12-item questionnaire that utilized self-reported physical work capacity to estimate peak metabolic equivalents (METs) and has been shown to be a valid measurement of functional capacity.
PROM 11:The Multidimensional Impact of Cancer Risk Assessment (MICRA) | 1 Week Post Genetic Test Results via BCTA
  A 25-item tool use to assess participants and the specific impact of result disclosure after genetic testing. The assessment administers 4 point Likert-type questions (never=0 to often=5) regarding how individuals feel after being told their genetic test results.
  Distress subscale = Items 1-4, 7 & 8; Uncertainty subscale = Items 9-12, 14-17 & 20; Positive experiences subscale (reverse scored) = Items 5, 6, 18 & 19. Subscales are scored by summing circled numbers
PROM 12: The Knowgene | 1 Week Post Genetic Test Results via BCTA
  The number of participants and their general cancer genetic knowledge after cancer genetic counseling and multigene panel testing.
PROM 13: Breast Cancer Treatment Application Review Survey (BCTA) | 12-months Post-Enrollment
  Patient satisfaction with the app will be measured by utilizing the Breast Cancer Treatment Application Review Survey. The survey will be administered to participants using the application at the 12-month mark, to better understand any barriers to using the app and which aspects were most useful to patients. The 10 item assessment uses 5-point Likert-type questions (strongly disagree to strongly agree) to assess their experience on the application.
PROM 14: Functional Assessment Of Cancer Therapy-Endocrine Subscale (FACT-ES) Score | 2 to 3 Months Post Start of Endocrine Treatment via Breast Cancer Treatment App
  Investigators will measure relative changes in adverse symptom burden using the Functional Assessment Of Cancer Therapy-Endocrine Subscale (FACT-ES) questionnaire. The FACT-ES is a 46-item questionnaire asking participants to report how much they have been impacted by a variety of symptoms on a 5-point scale where 0 = not at all and 4 = very much. Total raw scores range from 0 to 184, with higher scores indicating greater impact from symptoms.
PROM 15: System-Usability Score (SUS) | 12-months Post-Enrollment
  Usability will be assessed using the System Usability Scale (SUS). We wil collect the input of breast cancer patients to the SUS questions, using in-app surveys and will calculate the SUS score. We will assess overall satisfaction with the app by asking users to provide an answer to the question "How likely are you to recommend this product to a friend" on a scale of 0-10.
PROM 16: Distress Thermometer | At baseline, 6 months and 12 months after enrollment
  Participants will be asked to rate their level of distress over the past week on a scale from 0 to 10, where 0 represents no distress and 10 represents extreme distress.
PROM 17: Post Operative Questionnaires | 1 to 10 days after surgery
  Post-operative measures at one to 10 days after surgery, as assessed by our study-specific post-operative survey. This survey will ask patients on the app to report and rate symptoms that they may experience after surgery, including pain, numbness, fever, shortness of breath, tenderness around the incision site, fatigue, and anxiety.
Visits to the Breast Clinic | 3, 9 and 15 months after enrollment
  Number of visits to the breast clinic, as captured by auditing our booking system.
Phone Calls and Emails to the Breast Clinic | 3, 6, and 15 months after enrollment
  Number of calls and emails to the breast clinic, as captured by auditing the breast triage line and email.
Emergency Department Visits | 15 months post enrollment
  The number of emergency department visits recorded in the National Ambulatory Care Reporting System (NACRS) among ABODE study participants.
Unplanned Hospital Admissions | 15 months post enrollment
  The number of unplanned hospital admissions recorded in NACRS for ABODE study participants.
Outpatient Clinic Visits | 15 months post enrollment
  The number of outpatient clinic visits documented in NACRS among ABODE study participants.
Physical Activity Level (Steps per Day) | 13 months after enrollment (whole duration of the study)
  Daily step count recorded via Fitbit to assess trends in physical activity levels among study participants. Days without Fitbit data will be excluded from analysis.
Exercise Heart Rate | 13 months after enrollment (whole duration of the study)
  Average heart rate recorded during exercise sessions as measured by Fitbit, providing insights into cardiovascular response and fitness levels among study participants. Days without Fitbit data will be excluded from analysis.
Sleep Duration | 13 months after enrollment (whole duration of the study)
  Total sleep duration (in hours) per night as recorded by Fitbit, providing insight into distress levels that may affect sleep quality. Days without Fitbit data will be excluded.
Hospital Admissions | 15 months post enrollment
  The number of hospital admissions recorded in the Discharge Abstract Database (DAD) among ABODE study participants.
Length of Hospital Stay | 15 months post enrollment
  Total number of days spent in the hospital per admission, as recorded in the DAD, to assess the duration of inpatient care.
Discharge Outcomes | 15 months post enrollment
  The type of discharge (e.g., home, rehabilitation facility, or readmission) recorded in the DAD, providing insights into patient recovery.
Post-Surgical Complications | 15 months post enrollment
  The number of post-surgical complications (e.g., infections, readmissions due to complications) recorded in the DAD, contributing to the assessment of patient recovery.
Wait Times | 15 months post enrolment
  The length of time from referral to procedure or discharge, as recorded in the Wait Times Information System (TIS), which tracks wait times for surgeries, diagnostic imaging (e.g., MRI, CT), and alternate level of care (ALC) in Ontario hospitals. This measure will assess differences in wait times between study groups, offering insight into system efficiency and access to care.

CONTACTS AND LOCATIONS:
Overall Officials: Tulin Cil, MD, MEd, Principal Investigator — University Health Network, Toronto
Locations (1):
- Tulin Cil, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mac A, Kalia M, Reel E, Amir E, Isenberg A, Kim RH, Kennedy E, Koch CA, Li M, McCready D, Metcalfe K, Okrainec A, Papadakos J, Rotstein S, Rodin G, Xu W, Zhong T; ABODE Study Group; Cil TD. At-home Breast Oncology care Delivered with EHealth solutions (ABODE) study protocol: a randomised controlled trial. BMJ Open. 2025 May 8;15(5):e091579. doi: 10.1136/bmjopen-2024-091579. PMID 40345693